CLINICAL TRIAL: NCT03116113
Title: A Dose Escalation (Phase 1), and Dose Expansion (Phase 2/3) Clinical Trial of Retinal Gene Therapy for X-linked Retinitis Pigmentosa Using an Adeno-Associated Viral Vector (AAV8) Encoding Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: A Clinical Trial of Retinal Gene Therapy for X-linked Retinitis Pigmentosa Using BIIB112
Acronym: XIRIUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 274RP101; 2016-003852-60 (EudraCT Number)
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; Ophthalmology; Gene Therapy; Retinitis Pigmentosa GTPase Regulator (RPGR); AAV8
MeSH Terms: conditions — Cone-Rod Dystrophy, X-Linked, Type 1 | interventions — Cotoretigene Toliparvovec

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: BIIB112 Dose 1 (Experimental): Participants will receive a single Dose 1 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 1: BIIB112 Dose 2 (Experimental): Participants will receive a single Dose 2 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 1: BIIB112 Dose 3 (Experimental): Participants will receive a single Dose 3 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 1: BIIB112 Dose 4 (Experimental): Participants will receive a single Dose 4 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 1: BIIB112 Dose 5 (Experimental): Participants will receive a single Dose 5 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 1: BIIB112 Dose 6 (Experimental): Participants will receive a single Dose 6 of BIIB112 by sub-retinal injection on Day 0.
  Interventions: Biological: BIIB112
- Part 2: BIIB112 High Dose (Experimental): Participants will receive a single high dose of BIIB112 by sub-retinal injection.
  Interventions: Biological: BIIB112
- Part 2: BIIB112 Low Dose (Experimental): Participants will receive a single low dose of BIIB112 by sub-retinal injection.
  Interventions: Biological: BIIB112
- Part 2: Untreated Group (No Intervention): Participants will receive no intervention to allow for a controlled comparison.

INTERVENTIONS:
Biological: BIIB112 — Administered as specified in the treatment arm.
  Other Names: AAV8-RPGR
  Arms: Part 1: BIIB112 Dose 1; Part 1: BIIB112 Dose 2; Part 1: BIIB112 Dose 3; Part 1: BIIB112 Dose 4; Part 1: BIIB112 Dose 5; Part 1: BIIB112 Dose 6; Part 2: BIIB112 High Dose; Part 2: BIIB112 Low Dose

SUMMARY:
The objective of the study is to evaluate the safety, tolerability and efficacy of a single sub-retinal injection of BIIB112 in participants with X-linked retinitis pigmentosa (XLRP).

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

Part 1:

* Participants with genetically confirmed diagnosis of XLRP (with RPGR mutation).
* Participant with active disease clinically visible within the macular region in both eyes.

Part 2:

- Participant with mean total retinal sensitivity in the study eye as assessed by microperimetry ≥ 0.1 dB and ≤8 dB.

Key exclusion Criteria:

Parts 1 and 2:

* Participant with history of amblyopia in either eye.
* Participated in a gene therapy trial previously or a clinical trial with an investigational drug in the past 12 weeks or received a gene/cell-based therapy at any time previously.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- United States (5):
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
- United Kingdom (3):
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Result] Cehajic-Kapetanovic J, Xue K, Martinez-Fernandez de la Camara C, Nanda A, Davies A, Wood LJ, Salvetti AP, Fischer MD, Aylward JW, Barnard AR, Jolly JK, Luo E, Lujan BJ, Ong T, Girach A, Black GCM, Gregori NZ, Davis JL, Rosa PR, Lotery AJ, Lam BL, Stanga PE, MacLaren RE. Initial results from a first-in-human gene therapy trial on X-linked retinitis pigmentosa caused by mutations in RPGR. Nat Med. 2020 Mar;26(3):354-359. doi: 10.1038/s41591-020-0763-1. Epub 2020 Feb 24. PMID 32094925
- [Derived] Raji S, Taylor LJ, Josan AS, MacLaren RE, Cehajic-Kapetanovic J. Early-Onset Cone Photoreceptor Degeneration Is Associated With High Myopia in RPGR-Related Retinal Dystrophy. J Ophthalmol. 2025 Jun 11;2025:4244740. doi: 10.1155/joph/4244740. eCollection 2025. PMID 40535564
- [Derived] Lam BL, Pennesi ME, Kay CN, Panda S, Gow JA, Zhao G, MacLaren RE; XIRIUS Study Group. Assessment of Visual Function with Cotoretigene Toliparvovec in X-Linked Retinitis Pigmentosa in the Randomized XIRIUS Phase 2/3 Study. Ophthalmology. 2024 Sep;131(9):1083-1093. doi: 10.1016/j.ophtha.2024.02.023. Epub 2024 Feb 28. PMID 38423215
- [Derived] von Krusenstiern L, Liu J, Liao E, Gow JA, Chen G, Ong T, Lotery AJ, Jalil A, Lam BL, MacLaren RE; XIRIUS Part 1 Study GroupXOLARIS Study Group. Changes in Retinal Sensitivity Associated With Cotoretigene Toliparvovec in X-Linked Retinitis Pigmentosa With RPGR Gene Variations. JAMA Ophthalmol. 2023 Mar 1;141(3):275-283. doi: 10.1001/jamaophthalmol.2022.6254. PMID 36757689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at investigational sites in the United Kingdom (UK) and the United States (US) from 08 March 2017 to 18 November 2020.
Pre-assignment Details: A total of 50 participants with X-Linked Retinitis Pigmentosa (XLRP) were enrolled in the study (18 participants in Part 1 and 32 participants in Part 2). Of these, 47 participants completed the study (18 participants in Part 1 and 29 in Part 2).
Groups:
- Part 1: BIIB112 Dose 1: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 1 (5 × 10^9 vector genomes {vg} ) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 1: BIIB112 Dose 2: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 2 (1 × 10^10 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 1: BIIB112 Dose 3: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 3 (5 × 10^10 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 1: BIIB112 Dose 4: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 4 (1 × 10^11 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 1: BIIB112 Dose 5: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 5 (2.5 × 10^11 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 1: BIIB112 Dose 6: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 6 (5 × 10^11 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 2: Untreated Group: Participants received no intervention to allow for a controlled comparison.
- Part 2: BIIB112 Low Dose: Followed by vitrectomy and retinal detachment in study eye, participants received a single low dose (5 × 10^10 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 2: BIIB112 High Dose: Followed by vitrectomy and retinal detachment in study eye, participants received a single high dose (2.5 × 10^11 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
Period: Part 1 (Day 0 up to Month 24)
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6 | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Month 25 up to Month 36)
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6 | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 11 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrew due to Coronavirus 2019COVID-19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Groups:
- Part 1: BIIB112 Dose 1: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 1 (5 × 10^9 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Total: Total of all reporting groups
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6 | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 11 | 12 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (6.35) | 34.3 (10.69) | 30.0 (2.65) | 33.3 (14.57) | 25.0 (5.00) | 32.3 (15.31) | 33.7 (13.83) | 30.6 (8.83) | 26.8 (7.11) | 30.7 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 11 | 12 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 5 | 11
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 2 | 7 | 8 | 7 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: White | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 9 | 12 | 45
  Race: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs are defined as any of the following events considered to be related to study drug: Sustained decrease in best-corrected visual acuity (BCVA) of ≥30 letters on the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart compared to baseline (sustained is defined as lasting 48 hours or more until recovery, with recovery defined as visual acuity (VA) returning to within 10 letters of baseline VA. An exception is made for surgery-related events occurring in close temporal association {within <24 hours} of the surgery); Vitreous inflammation, vitritis (>Grade 3 using standardized Nussenblatt vitreous inflammation scale grading); Any clinically significant retinal damage observed that is not directly attributed to complications of surgery; Any clinically relevant suspected unexpected serious adverse reaction, with the exception of vision loss or vision threatening.
Time Frame: Up to Month 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are defined as the AEs starting or worsening on or after the day of the first surgery.
Time Frame: Day 0 (surgery) in Part 1 of the study up to 24 months
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Participants | 3 | 3 | 3 | 3 | 3 | 3

3. Primary Outcome: Part 2: Percentage of Study Eyes With ≥7 Decibels (dB) Improvement From Baseline at ≥5 Points Out of the 16 Central Loci Points of the 10-2 Grid Assessed by Macular Integrity Assessment (MAIA) Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0', or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Improvement in Retinal Sensitivity in center grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points out of the 16 central points.
Time Frame: Month 12
Population: Intent-to-treat (ITT) analysis set included all participants that were randomized under the 3-arm randomization schedules. "Overall number of participants analyzed" signifies the number of participants with data available for analysis of this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of study eyes
Units Other Than Participants: Study eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 8 | 8
Number analyzed (Study eyes) | 9 | 8 | 8
percentage of study eyes | 22.2 [6.1 to 49.0] | 37.5 [14.7 to 65.5] | 25.0 [6.9 to 53.8]
Statistical Analysis 1: Comparison: Part 2: Untreated Group vs Part 2: BIIB112 Low Dose; Test type: Superiority; p = 0.3181, Fisher's Exact-Boschloo test
Statistical Analysis 2: Comparison: Part 2: Untreated Group vs Part 2: BIIB112 High Dose; Test type: Superiority; p = 0.5177, Fisher's Exact-Boschloo test

4. Primary Outcome: Part 2: Number of Participants With TEAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are defined as AEs starting on or after the day of the first surgery.
Time Frame: Day 0 (surgery) in Part 2 of the study up to 12 months
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 11 | 12
Participants | 5 | 11 | 12

5. Secondary Outcome: Part 1: Percentage of Study Eyes With ≥7 dB Improvement From Baseline at ≥5 Points Out of the 16 Central Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Improvement in Retinal Sensitivity in center grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points out of the 16 central points.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112). 'Overall number of participants analyzed' signifies the number of participants with data available for analysis of outcome measure. 'Number of participants analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of study eyes
Units Other Than Participants: study eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3
Number analyzed (study eyes) | 3 | 2 | 3 | 3 | 3 | 3
percentage of study eyes
  Month 1 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 9 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 12: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Month 12: number analyzed (study eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Month 12 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6]
  Month 18: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Month 18: number analyzed (study eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Month 18 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2]
  Month 24: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Month 24: number analyzed (study eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Month 24 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

6. Secondary Outcome: Part 1: Percentage of Study Eyes With ≥7 dB Improvement From Baseline at ≥5 Points Out of the 68 Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Improvement in Retinal Sensitivity in whole grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points of the grid as a whole (68 points).
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of study eyes
Units Other Than Participants: study eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3
Number analyzed (study eyes) | 3 | 2 | 3 | 3 | 3 | 3
percentage of study eyes
  Month 1 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 6 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0]
  Month 9 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 12: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Month 12: number analyzed (study eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Month 12 | 0.0 [0.0 to 70.8] | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2]
  Month 18: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Month 18: number analyzed (study eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Month 18 | 0.0 [0.0 to 70.8] | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 50.0 [1.3 to 98.7]
  Month 24: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Month 24: number analyzed (study eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Month 24 | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 99.2]

7. Secondary Outcome: Part 1: Change From Baseline in Mean Sensitivity of the 16 Central Loci Points Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' is assigned a value of '-1' by MAIA in the calculation. Improvement in mean sensitivity in center grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points out of the 16 central points. Here negative values indicate a decline in retinal sensitivity.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 4 | 6 | 6 | 6 | 6
dBs
  Baseline: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Baseline: Study Eye | 0.33 (1.748) | 1.78 (1.282) | 3.35 (0.911) | 6.52 (3.398) | 13.46 (6.316) | 7.75 (7.742)
  Baseline: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Baseline: Non-Study Eye | 0.23 (1.358) | 3.31 (2.563) | 6.92 (2.221) | 8.21 (5.570) | 13.71 (8.447) | 7.54 (7.542)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye | 0.52 (0.477) | -0.09 (0.928) | 6.10 (0.844) | 1.19 (6.094) | -0.63 (4.154) | -1.90 (7.686)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye | 0.42 (1.122) | -0.81 (1.768) | -0.98 (1.531) | -0.19 (0.272) | 1.40 (2.690) | 0.19 (2.063)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye | 0.40 (0.407) | 0.47 (1.282) | 5.63 (2.394) | 1.73 (8.714) | -3.58 (7.476) | -3.35 (2.894)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye | -0.06 (0.534) | -0.91 (0.575) | -1.15 (2.094) | 0.33 (1.134) | 2.06 (1.137) | -0.42 (0.289)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye | 0.54 (0.485) | -0.06 (0.265) | 5.10 (1.890) | 3.25 (8.199) | -2.38 (5.177) | 0.85 (5.105)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Non-Study Eye | -0.17 (0.344) | -0.34 (2.607) | -1.19 (1.535) | 2.10 (3.437) | 2.19 (0.933) | -0.65 (1.156)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye | 0.21 (0.219) | 0.09 (1.282) | 4.65 (3.851) | 3.69 (6.308) | -2.50 (5.314) | 0.77 (7.096)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Non-Study Eye | -0.35 (0.509) | 0.19 (2.210) | 0.20 (2.751) | -0.06 (1.789) | 2.52 (1.714) | 0.40 (2.032)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Study Eye | 0.19 (0.272) | 0.13 (1.945) | 4.10 (2.908) | 3.98 (5.090) | 2.25 (2.121) | 0.56 (5.590)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Non-Study Eye | -0.10 (0.355) | -1.09 (1.370) | -1.02 (0.581) | 0.42 (1.951) | 2.31 (2.990) | -0.29 (1.835)
  Change From Baseline at Month 18: Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Study Eye | 0.21 (0.473) | -1.13 (0.177) | 2.69 (2.507) | 2.92 (5.550) | -2.79 (6.733) | -1.09 (5.436)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Non-Study Eye | -0.33 (0.577) | -1.09 (1.282) | 0.02 (0.940) | -0.67 (0.806) | 1.92 (3.085) | -0.59 (2.607)
  Change From Baseline at Month 24: Study Eye: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | 0.04 (0.253) | -1.88 (NA) — Standard deviation (SD) cannot be estimated for 1 participant. | 2.75 (2.683) | 1.48 (5.236) | -4.90 (5.250) | -1.88 (5.862)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -0.46 (0.469) | -1.63 (NA) — SD cannot be estimated for 1 participant. | -0.33 (1.347) | -0.56 (1.207) | 0.71 (3.263) | -2.19 (2.189)

8. Secondary Outcome: Part 1: Change From Baseline in Mean Sensitivity of the 68 Central Loci Points Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' is assigned a value of '-1' by MAIA in the calculation. Improvement in mean sensitivity in whole grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points of the grid as a whole (68 points). Here negative values indicate a decline in retinal sensitivity.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 4 | 6 | 6 | 6 | 6
dBs
  Baseline: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Baseline: Study Eye | -0.19 (0.690) | 0.20 (0.281) | 0.21 (0.435) | 2.22 (1.536) | 8.87 (10.784) | 4.26 (6.732)
  Baseline: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Baseline: Non-Study Eye | -0.38 (0.540) | 1.47 (1.061) | 1.50 (1.419) | 2.30 (1.559) | 9.11 (12.466) | 5.35 (8.579)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye | 0.12 (0.309) | 0.24 (1.185) | 2.42 (0.283) | 0.08 (2.436) | 0.56 (3.243) | -1.69 (4.341)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye | 0.18 (0.481) | -0.76 (1.165) | -0.08 (0.938) | -0.11 (0.111) | 1.24 (1.639) | -0.66 (1.474)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye | 0.14 (0.137) | 0.74 (1.820) | 2.44 (1.564) | 0.58 (5.061) | -1.87 (4.073) | -0.60 (1.383)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye | -0.06 (0.292) | -0.29 (1.549) | -0.29 (1.351) | 0.68 (1.223) | 1.38 (1.005) | -0.65 (0.407)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye | 0.04 (0.334) | 0.19 (0.957) | 2.28 (1.534) | 0.90 (5.011) | -0.60 (1.596) | 0.51 (2.154)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Non-Study Eye | -0.24 (0.331) | -0.32 (1.872) | -0.51 (0.773) | 3.86 (5.648) | 1.76 (0.470) | -0.84 (1.101)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye | -0.18 (0.145) | 0.31 (1.456) | 2.02 (2.177) | 0.90 (4.233) | -0.87 (2.229) | -0.13 (4.044)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Non-Study Eye | -0.37 (0.467) | -0.12 (1.830) | 1.66 (1.790) | 0.77 (1.405) | 2.05 (0.816) | -0.41 (1.157)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Study Eye | -0.16 (0.165) | 0.30 (1.612) | 1.72 (1.892) | 1.28 (3.541) | -0.22 (2.600) | -0.41 (4.208)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 2 | 3
  Change From Baseline at Month 12: Non-Study Eye | -0.30 (0.417) | -0.46 (1.633) | -0.24 (0.153) | 0.76 (1.345) | 1.72 (1.144) | -0.82 (1.248)
  Change From Baseline at Month 18: Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Study Eye | -0.23 (0.213) | -0.50 (0.458) | 1.16 (1.144) | 1.37 (4.233) | -0.72 (1.253) | -1.32 (4.721)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 2 | 3 | 3 | 3 | 2
  Change From Baseline at Month 18: Non-Study Eye | -0.33 (0.412) | -0.57 (1.435) | 0.07 (0.509) | 0.18 (0.191) | 1.24 (1.265) | -1.19 (2.267)
  Change From Baseline at Month 24: Study Eye: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | -0.40 (0.382) | -0.96 (NA) — SD cannot be estimated for 1 participant. | 1.17 (1.190) | 0.98 (3.510) | -2.37 (1.225) | -2.26 (6.009)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 1 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -0.37 (0.427) | -1.44 (NA) — SD cannot be estimated for 1 participant. | 0.14 (0.221) | 0.24 (0.153) | 0.75 (1.427) | -1.73 (2.481)

9. Secondary Outcome: Part 1: Change From Baseline in Mean Best Corrected Visual Acuity (BCVA) Reported as Letters
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. BCVA was reported as number of letters read correctly by the participants using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate decline in BCVA.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
letters
  Baseline: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Study Eye | 27.67 (8.145) | 49.67 (9.452) | 64.33 (7.095) | 63.67 (20.551) | 70.67 (4.163) | 67.33 (15.044)
  Baseline: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Non-Study Eye | 60.67 (2.082) | 57.33 (5.686) | 66.33 (2.517) | 62.67 (22.279) | 73.33 (4.163) | 75.00 (4.583)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye | 3.67 (3.055) | 0.33 (2.517) | -1.00 (1.732) | -1.33 (6.506) | -0.67 (4.041) | -0.67 (10.693)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye | 3.00 (3.000) | 1.00 (4.359) | 1.00 (1.000) | 0.33 (0.577) | 2.00 (4.583) | -2.67 (1.155)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye | 6.33 (2.309) | 0.00 (3.606) | 0.67 (2.082) | 1.67 (4.726) | 0.33 (6.028) | 0.67 (6.506)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye | 3.00 (1.000) | 1.67 (1.528) | -1.67 (1.528) | 2.33 (2.309) | 4.67 (4.509) | -0.33 (0.577)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye | 5.00 (1.000) | -3.67 (3.786) | 0.33 (0.577) | 3.67 (5.686) | -3.67 (8.737) | -0.67 (5.033)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Non-Study Eye | -1.00 (7.211) | -0.67 (4.726) | -0.33 (3.215) | 3.67 (3.055) | 4.00 (4.359) | -0.67 (1.528)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye | 1.33 (4.619) | -0.67 (0.577) | 1.33 (4.509) | 4.00 (5.292) | -3.67 (16.073) | -2.33 (9.074)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Non-Study Eye | -5.00 (5.292) | -0.67 (5.033) | 1.00 (1.000) | 3.00 (3.606) | 5.67 (8.622) | 2.00 (4.359)
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Study Eye | 4.67 (4.509) | -2.00 (3.464) | 0.67 (5.132) | 4.33 (4.933) | -15.00 (40.286) | -2.33 (8.327)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye | -1.67 (2.309) | -0.33 (3.215) | -0.33 (0.577) | 2.00 (4.359) | 6.67 (6.429) | 1.00 (2.000)
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 18: Study Eye | 3.00 (8.718) | -2.00 (3.606) | -3.33 (5.132) | 3.33 (3.786) | -9.33 (28.919) | -5.00 (8.544)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye | -4.00 (6.245) | 0.00 (5.000) | -0.33 (2.517) | 1.33 (2.517) | 5.00 (7.810) | -0.33 (5.508)
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | -2.00 (15.588) | -2.00 (5.292) | -3.33 (3.215) | 5.00 (7.000) | -13.33 (32.747) | -5.67 (6.110)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -3.67 (5.508) | 0.67 (0.577) | -2.33 (1.528) | 2.33 (4.509) | 2.00 (7.810) | -2.00 (3.000)

10. Secondary Outcome: Part 1: Change From Baseline in Mean Low Luminance Visual Acuity (LLVA) Reported as Letters
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. LLVA was reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate decline in LLVA.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112). 'Overall number of participants analyzed' signifies the number of participants with data available for analysis of outcome measure.
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
letters
  Baseline: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Baseline: Study Eye |  |  | 41.00 (18.385) | 34.33 (29.939) | 58.00 (3.000) | 41.67 (34.646)
  Baseline: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Baseline: Non-Study Eye |  |  | 37.50 (24.749) | 37.67 (32.808) | 61.00 (2.646) | 57.33 (14.844)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye |  |  | 10.00 (9.899) | 0.33 (0.577) | 3.00 (5.292) | 4.67 (26.502)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye |  |  | 10.00 (18.385) | -0.33 (7.506) | 3.00 (5.196) | -4.33 (7.572)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye |  |  | 14.00 (11.314) | 7.33 (6.658) | -14.33 (38.214) | -7.67 (10.263)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye |  |  | 10.00 (16.971) | 1.00 (1.000) | 3.00 (4.583) | 2.00 (3.464)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye |  |  | 11.50 (7.778) | 8.33 (7.234) | -16.67 (35.810) | 7.33 (9.713)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 6: Non-Study Eye |  |  | 8.00 (15.556) | 1.67 (2.887) | 5.33 (1.155) | 0.67 (3.215)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye |  |  | 0.50 (4.950) | 10.00 (6.557) | -14.33 (37.820) | 4.33 (8.083)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 9: Non-Study Eye |  |  | 0.50 (4.950) | 2.00 (4.359) | 2.00 (3.464) | 3.33 (2.309)
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 12: Study Eye |  |  | 3.50 (0.707) | 16.00 (13.454) | -11.33 (40.612) | 8.33 (11.590)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye |  |  | 7.00 (9.899) | 6.67 (8.327) | 9.00 (4.359) | 4.00 (6.083)
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 18: Study Eye |  |  | 6.50 (7.778) | 10.67 (8.622) | -12.33 (40.079) | 8.33 (5.508)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye |  |  | 9.00 (21.213) | 2.33 (2.517) | 5.67 (4.726) | -4.33 (7.234)
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye |  |  | 3.00 (8.485) | 9.33 (14.295) | -14.67 (38.371) | -1.67 (6.506)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye |  |  | 5.50 (24.749) | 0.67 (4.041) | 3.33 (3.512) | -12.67 (11.547)

11. Secondary Outcome: Part 1: Percentage of Eyes With a ≥15 Letters Increase From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥15 letters increase from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

12. Secondary Outcome: Part 1: Percentage of Eyes With a ≥15 Letters Increase From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥15 letters increase from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

13. Secondary Outcome: Part 1: Percentage of Eyes With a ≥10 Letters Increase From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥10 letters increase from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]

14. Secondary Outcome: Part 1: Percentage of Eyes With a ≥10 Letters Increase From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥10 letters increase from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

15. Secondary Outcome: Part 1: Percentage of Eyes With a ≥5 Letters Increase From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥5 letters increase from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.03 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]

16. Secondary Outcome: Part 1: Percentage of Eyes With a ≥5 Letters Increase From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥5 letters increase from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 100.0 [15.8 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 100.0 [15.8 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 50.0 [1.3 to 98.7] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]

17. Secondary Outcome: Part 1: Percentage of Eyes With a ≥15 Letters Loss From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥15 letters loss from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

18. Secondary Outcome: Part 1: Percentage of Eyes With a ≥15 Letters Loss From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥15 letters loss from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 2
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 2
  Month 1: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 3
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 2 | 3 | 3
  Month 3: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]

19. Secondary Outcome: Part 1: Percentage of Eyes With a ≥10 Letters Loss From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥10 letters loss from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

20. Secondary Outcome: Part 1: Percentage of Eyes With a ≥10 Letters Loss From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥10 letters loss from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]

21. Secondary Outcome: Part 1: Percentage of Eyes With a ≥5 Letters Loss From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥5 letters loss from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 66.7 [9.4 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 33.3 [0.8 to 99.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]

22. Secondary Outcome: Part 1: Percentage of Eyes With a ≥5 Letters Loss From Baseline for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a ≥5 letters loss from baseline for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.00 [0.0 to 70.8] | 33.3 [0.8 to 90.6]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 100.0 [29.2 to 100.0]

23. Secondary Outcome: Part 1: Percentage of Eyes With Change From Baseline > -5 Letters for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Percentage of eyes with a change from baseline of ≥ -5 letters for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112).
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 1: Non-Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 3: Non-Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Study Eye | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 6: Non-Study Eye | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 9: Non-Study Eye | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 12: Non-Study Eye | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Study Eye | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 18: Non-Study Eye | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2]
  Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Study Eye | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Month 24: Non-Study Eye | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2]

24. Secondary Outcome: Part 1: Percentage of Eyes With Change From Baseline > -5 Letters for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Percentage of eyes with a change from baseline of ≥ -5 letters for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 3
Number analyzed (eyes) | 0 | 0 | 4 | 6 | 6 | 6
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 1: Non-Study Eye |  |  | 100.0 [15.8 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2]
  Month 3: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  Month 3: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 3: Non-Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0]
  Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 6: Non-Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 9: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0]
  Month 9: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 9: Non-Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 12: Non-Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Month 18: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0]
  Month 18: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 18: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 33.3 [0.8 to 90.6]
  Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Study Eye |  |  | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2]
  Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 2 | 3 | 3 | 3
  Month 24: Non-Study Eye |  |  | 50.0 [1.3 to 98.7] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 70.8]

25. Secondary Outcome: Part 1: Change From Baseline in Central Ellipsoid Area
Description: Spectral Domain Optical Coherence Tomography (SD-OCT) was used to assess change in central ellipsoid area. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates a decline in central ellipsoid area.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112). 'Number analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: square millimeters (mm^2)
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
square millimeters (mm^2)
  Baseline: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Study Eye | 0.140 (0.1637) | 2.750 (4.7631) | 0.137 (0.1582) | 0.193 (0.1686) | 8.327 (13.8600) | 3.107 (5.2001)
  Baseline: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Baseline: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Baseline: Non-Study Eye | 0.130 (0.0985) | 2.313 (3.7500) | 0.093 (0.0814) | 0.465 (0.1061) | 14.307 (24.1914) | 5.257 (8.8720)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye | -0.077 (0.1159) | -0.493 (0.8545) | -0.103 (0.1050) | -0.050 (0.0458) | -1.360 (2.2863) | -1.310 (2.2258)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye | -0.060 (0.0265) | -0.383 (0.4508) | -0.020 (0.0693) | -0.080 (0.0566) | -0.410 (0.7645) | 0.873 (1.5824)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 2 | 3
  Change From Baseline at Month 3: Study Eye | -0.100 (0.1249) | -0.560 (0.9699) | -0.110 (0.1153) | -0.060 (0.0529) | -2.255 (3.0335) | -2.960 (5.0319)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 3: Non-Study Eye | -0.093 (0.0404) | -0.407 (0.4895) | -0.043 (0.0379) | -0.095 (0.0495) | -0.407 (0.7778) | -0.040 (0.0566)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 2
  Change From Baseline at Month 6: Study Eye | -0.120 (0.1375) | -0.527 (0.9122) | -0.113 (0.1206) | -0.070 (0.0624) | -4.847 (8.1176) | -0.055 (0.0778)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 6: Non-Study Eye | -0.093 (0.0404) | -0.410 (0.4951) | -0.060 (0.0529) | -0.120 (0.0424) | -0.983 (1.7747) | -0.050 (0.0707)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye | -0.127 (0.1419) | -0.540 (0.9353) | -0.117 (0.1258) | -0.063 (0.0551) | -5.640 (9.4830) | -2.960 (5.0664)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 9: Non-Study Eye | -0.097 (0.0451) | -0.437 (0.5326) | -0.063 (0.0569) | -0.120 (0.0141) | -1.100 (1.9504) | -0.050 (0.0707)
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Study Eye | -0.130 (0.1473) | -0.560 (0.9699) | -0.117 (0.1258) | -0.053 (0.0551) | -5.623 (9.4975) | -3.007 (5.1386)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye | -0.097 (0.0451) | -0.447 (0.5353) | -0.033 (0.1266) | -0.120 (0.0424) | -1.010 (2.0313) | 0.997 (1.8312)
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 18: Study Eye | -0.133 (0.1528) | -0.567 (0.9815) | -0.137 (0.1582) | 0.027 (0.1617) | -5.633 (9.4975) | -2.993 (5.1155)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye | 0.1528 (0.0709) | -0.450 (0.5408) | -0.027 (0.1201) | -0.115 (0.0919) | -1.107 (2.0124) | 0.590 (1.1364)
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | -0.133 (0.1528) | -0.573 (0.9930) | -0.137 (0.1582) | 0.010 (0.1552) | -5.657 (9.5292) | -3.010 (5.1357)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -0.117 (0.0764) | -0.443 (0.5297) | -0.060 (0.0794) | -0.150 (0.0283) | -1.163 (2.0063) | 0.367 (0.7505)

26. Secondary Outcome: Part 1: Change From Baseline in Central Horizontal Ellipsoid Width
Description: SD-OCT was used to assess change in central horizontal ellipsoid width. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates a decline in central horizontal ellipsoid width.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Microns
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
Microns
  Baseline: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Study Eye | 162.67 (175.104) | 1375.33 (2382.147) | 248.00 (275.158) | 462.33 (400.775) | 2411.33 (3048.253) | 745.67 (774.448)
  Baseline: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Baseline: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Baseline: Non-Study Eye | 355.67 (378) | 1383.67 (396.581) | 250.00 (33.139) | 792.00 (300.409) | 3341.00 (4556.473) | 937.67 (1088.262)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 1: Study Eye | -56.33 (73.894) | -311.00 (538.668) | -174.00 (162.567) | -26.33 (24.007) | 4556.473 (248.605) | 88.67 (422.044)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 1: Non-Study Eye | -62.33 (40.216) | -321.67 (557.143) | 47.33 (226.509) | -56.00 (63.640) | -14.00 (113.331) | 977.33 (1814.500)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye | -73.00 (70.193) | -318.00 (550.792) | -174.33 (163.022) | -89.33 (125.644) | -369.00 (271.070) | -453.33 (554.795)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye | -149.00 (80.988) | -333.33 (577.350) | -60.67 (78.258) | -151.00 (15.556) | -19.00 (123.503) | 1008.33 (1869.924)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye | -115.67 (105.624) | -318.67 (551.947) | -175.67 (164.852) | -146.67 (129.454) | -1070.67 (1365.685) | -461.33 (553.453)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 6: Non-Study Eye | -158.67 (65.033) | -347.00 (601.022) | -76.33 (79.135) | -195.50 (6.364) | -20.00 (144.503) | -108.50 (153.442)
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 9: Study Eye | -127.00 (121.025) | -321.33 (556.566) | -178.33 (168.548) | -149.00 (131.936) | -1096.33 (1343.289) | -441.00 (505.720)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 2
  Change From Baseline at Month 9: Non-Study Eye | -175.00 (39.585) | -348.00 (602.754) | -77.33 (79.053) | -202.50 (4.950) | -81.67 (217.721) | -124.00 (175.362)
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Study Eye | -130.00 (125.300) | -238.33 (412.805) | -217.00 (225.980) | -106.33 (132.666) | -1055.33 (1394.128) | -463.00 (537.199)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye | -181.67 (30.665) | -349.33 (605.063) | -35.67 (255.895) | -113.50 (47.376) | -143.00 (221.007) | 1108.00 (2145.532)
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 18: Study Eye | -131.00 (126.740) | -239.33 (414.537) | -248.00 (275.158) | 21.67 (332.031) | -1059.67 (1438.362) | -461.67 (530.381)
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 18: Non-Study Eye | -316.67 (213.601) | -354.67 (614.301) | -168.67 (161.122) | -188.00 (65.054) | -113.00 (242.736) | 1078.67 (2094.819)
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | -131.33 (127.222) | -242.33 (419.734) | -248.00 (275.158) | -43.33 (243.904) | -1162.00 (1352.050) | -465.67 (587.699)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 2 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -329.33 (235.434) | -358.00 (620.074) | -145.67 (162.543) | -254.50 (7.778) | -159.67 (265.038) | 1065.67 (2074.136)

27. Secondary Outcome: Part 1: Change From Baseline in Fundus Autofluoroscence- Mean Total Area of Preserved Autofluoroscence
Description: Fundus Autofluoroscence was used to assess the total area of preserved autofluoroscence. Areas of preserved AF were identified as well-demarcated regions of relative hyper autofluorescence (hyper AF) compared with the background areas of surrounding atrophy. A negative change from baseline indicates a decline in total area of preserved autofluoroscence.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: Safety analysis set included all participants who received study treatment (vitrectomy/BIIB112). 'Overall number of participants analyzed' signifies the number of participants with data available for analysis of outcome measure. 'Number analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
Number analyzed (eyes) | 2 | 0 | 2 | 0 | 0 | 0
mm^2
  Baseline: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: Study Eye | 27.050 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Baseline: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Baseline: Non-Study Eye | 22.910 (NA) — SD cannot be estimated for 1 participant. |  | 50.640 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 1: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 1: Study Eye | -1.820 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 1: Non-Study Eye | -2.420 (NA) — SD cannot be estimated for 1 participant. |  | -8.620 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 3: Study Eye | -2.940 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 3: Non-Study Eye | -2.650 (NA) — SD cannot be estimated for 1 participant. |  | -5.150 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 6: Study Eye | -3.460 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 6: Non-Study Eye | -3.050 (NA) — SD cannot be estimated for 1 participant. |  | -6.530 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 9: Study Eye | -3.470 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 9: Non-Study Eye | -3.100 (NA) — SD cannot be estimated for 1 participant. |  | -9.130 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 12: Study Eye | -3.640 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 12: Non-Study Eye | -3.760 (NA) — SD cannot be estimated for 1 participant. |  | -9.220 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 18: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 18: Study Eye | -3.670 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 1 | 0 | 0 | 0
  Change From Baseline at Month 18: Non-Study Eye | -3.830 (NA) — SD cannot be estimated for 1 participant. |  | -11.700 (NA) — SD cannot be estimated for 1 participant. |  |  |
  Change From Baseline at Month 24: Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 24: Study Eye | -3.740 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 1 | 0 | 0 | 0 | 0 | 0
  Change From Baseline at Month 24: Non-Study Eye | -4.120 (NA) — SD cannot be estimated for 1 participant. |  |  |  |  |

28. Secondary Outcome: Part 1: Change From Baseline in Fundus Autofluoroscence- Mean Distance From Foveal Center (FC) to Nearest Border of Preserved Autofluoroscence
Description: Fundus Autofluoroscence was used to assess the distance from FC to nearest border of preserved autofluoroscence. A negative change from baseline indicates a decline in the total area of preserved autofluoroscence.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 18, and 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1
Number analyzed (eyes) | 4 | 2 | 2 | 2 | 2 | 2
mm^2
  Baseline: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Baseline: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Baseline: Study Eye | 2394.50 (665.387) | -39.00 (NA) — SD cannot be estimated for 1 participant. | 3018.00 (NA) — SD cannot be estimated for 1 participant. | 361.00 (NA) — SD cannot be estimated for 1 participant. | 2853.00 (NA) — SD cannot be estimated for 1 participant. |
  Baseline: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 1
  Baseline: Non-Study Eye | 2609.00 (386.080) | -24.00 (NA) — SD cannot be estimated for 1 participant. | 3052.00 (NA) — SD cannot be estimated for 1 participant. | 369.00 (NA) — SD cannot be estimated for 1 participant. | 2816.00 (NA) — SD cannot be estimated for 1 participant. | 4047.00 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 1: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 1: Study Eye | -33.00 (5.657) | -14.00 (NA) — SD cannot be estimated for 1 participant. | -52.00 (NA) — SD cannot be estimated for 1 participant. | -14.00 (NA) — SD cannot be estimated for 1 participant. | -5.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 1
  Change From Baseline at Month 1: Non-Study Eye | -255.50 (297.692) | -19.00 (NA) — SD cannot be estimated for 1 participant. | -281.00 (NA) — SD cannot be estimated for 1 participant. | -18.00 (NA) — SD cannot be estimated for 1 participant. | -12.00 (NA) — SD cannot be estimated for 1 participant. | -3.00 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 3: Study Eye | -87.00 (24.042) | -16.00 (NA) — SD cannot be estimated for 1 participant. | -138.00 (NA) — SD cannot be estimated for 1 participant. | -89.00 (NA) — SD cannot be estimated for 1 participant. | -104.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 1
  Change From Baseline at Month 3: Non-Study Eye | -276.50 (324.562) | -30.00 (NA) — SD cannot be estimated for 1 participant. | -375.00 (NA) — SD cannot be estimated for 1 participant. | -22.00 (NA) — SD cannot be estimated for 1 participant. | -93.00 (NA) — SD cannot be estimated for 1 participant. | -21.00 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 6: Study Eye | -128.50 (54.447) | -24.00 (NA) — SD cannot be estimated for 1 participant. | -179.00 (NA) — SD cannot be estimated for 1 participant. | -93.00 (NA) — SD cannot be estimated for 1 participant. | -122.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 6: Non-Study Eye | -297.00 (349.311) | -41.00 (NA) — SD cannot be estimated for 1 participant. | -462.00 (NA) — SD cannot be estimated for 1 participant. | -36.00 (NA) — SD cannot be estimated for 1 participant. | -102.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 9: Study Eye | -140.00 (41.012) | -35.00 (NA) — SD cannot be estimated for 1 participant. | -281.00 (NA) — SD cannot be estimated for 1 participant. | -94.00 (NA) — SD cannot be estimated for 1 participant. | -140.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 9: Non-Study Eye | -310.50 (333.047) | -58.00 (NA) — SD cannot be estimated for 1 participant. | -413.00 (NA) — SD cannot be estimated for 1 participant. | -38.00 (NA) — SD cannot be estimated for 1 participant. | 92.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1 | 0
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 2 | 0 | 1 | 1 | 1 | 0
  Change From Baseline at Month 12: Study Eye | -1489.50 (1829.285) |  | -282.00 (NA) — SD cannot be estimated for 1 participant. | -101.00 (NA) — SD cannot be estimated for 1 participant. | -708.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1 | 0
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 2 | 0 | 1 | 1 | 1 | 0
  Change From Baseline at Month 12: Non-Study Eye | -353.50 (318.905) |  | -422.00 (NA) — SD cannot be estimated for 1 participant. | -39.00 (NA) — SD cannot be estimated for 1 participant. | 89.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 18: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 18: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 18: Study Eye | -1493.00 (1829.992) | -55.00 (NA) — SD cannot be estimated for 1 participant. | -310.00 (NA) — SD cannot be estimated for 1 participant. | -123.00 (NA) — SD cannot be estimated for 1 participant. | -1278.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 18: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 18: Non-Study Eye | -358.00 (318.198) | -86.00 (NA) — SD cannot be estimated for 1 participant. | -425.00 (NA) — SD cannot be estimated for 1 participant. | -11.00 (NA) — SD cannot be estimated for 1 participant. | 65.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 24: Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 24: Study Eye | -1501.00 (1820.093) | -69.00 (NA) — SD cannot be estimated for 1 participant. | -226.00 (NA) — SD cannot be estimated for 1 participant. | -125.00 (NA) — SD cannot be estimated for 1 participant. | -1293.00 (NA) — SD cannot be estimated for 1 participant. |
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 2 | 1 | 1 | 1 | 1 | 0
  Change From Baseline at Month 24: Non-Study Eye | -391.00 (301.227) | -91.00 (NA) — SD cannot be estimated for 1 participant. | -2646.00 (NA) — SD cannot be estimated for 1 participant. | -13.00 (NA) — SD cannot be estimated for 1 participant. | 62.00 (NA) — SD cannot be estimated for 1 participant. |

29. Secondary Outcome: Part 1: Change From Baseline in Mean Volume of 30-Degree Hill of Vision
Description: Visual field testing was performed to assess the volume of 30-degree hill vision, reported as dBs. Reliability Factor (RF)=number of false positive responses + number of false negative responses/number of false positive presentations + number of false negative presentations*100. If there are 0 responses, then RF value=0. RFpositive=number of false positive responses/number of false positive presentations*100. If RF≤ 20% measurement is considered reliable. If 20% < RF ≤ 25% and RFpositive ≤ 10% measurement is also considered reliable. Otherwise if 20% < RF ≤ 25% and RFpositive > 10%, or RF > 25%, measurement is not reliable. Only reliable measurements were included for analysis of this outcome measure. Here negative values indicate decline in volume of 30-degree hill vision.
Time Frame: Baseline, Months 6, 12, and 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
Number analyzed (eyes) | 0 | 0 | 0 | 0 | 2 | 2
dBs
  Baseline: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Baseline: Study Eye |  |  |  |  | 2.73 (NA) — SD cannot be estimated for 1 participant. | 5.07 (NA) — SD cannot be estimated for 1 participant.
  Baseline: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Baseline: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Baseline: Non-Study Eye |  |  |  |  |  | 5.17 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Study Eye |  |  |  |  |  | -2.14 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Non-Study Eye |  |  |  |  |  | -1.10 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Change From Baseline at Month 12: Study Eye |  |  |  |  | 0.33 (NA) — SD cannot be estimated for 1 participant. | -2.80 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 12: Non-Study Eye |  |  |  |  |  | -1.02 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Change From Baseline at Month 24: Study Eye |  |  |  |  | -1.89 (NA) — SD cannot be estimated for 1 participant. | -3.08 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 24: Non-Study Eye |  |  |  |  |  | -2.11 (NA) — SD cannot be estimated for 1 participant.

30. Secondary Outcome: Part 1: Change From Baseline in Mean Volume of Full Field Hill of Vision
Description: Visual field testing was performed to assess the volume of full field of hill vision, reported as dBs. RF =number of false positive responses + number of false negative responses/number of false positive presentations + number of false negative presentations*100. If there are 0 responses, then RF value=0. RFpositive=number of false positive responses/number of false positive presentations*100. If RF≤ 20% measurement is considered reliable. If 20% < RF ≤ 25% and RFpositive ≤ 10% measurement is also considered reliable. Otherwise if 20% < RF ≤ 25% and RFpositive > 10%, or RF > 25%, measurement is not reliable. Only reliable measurements were included for analysis of this outcome measure. Here negative values indicate decline in volume of 30-degree hill vision.
Time Frame: Baseline, Months 6, 12, and 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
Number analyzed (eyes) | 0 | 0 | 0 | 0 | 2 | 2
dBs
  Baseline: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Baseline: Study Eye |  |  |  |  | 15.77 (NA) — SD cannot be estimated for 1 participant. | 18.31 (NA) — SD cannot be estimated for 1 participant.
  Baseline: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Baseline: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Baseline: Non-Study Eye |  |  |  |  |  | 23.41 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Study Eye |  |  |  |  |  | -0.86 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 6: Non-Study Eye |  |  |  |  |  | -4.91 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Change From Baseline at Month 12: Study Eye |  |  |  |  | 1.29 (NA) — SD cannot be estimated for 1 participant. | -2.98 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 12: Non-Study Eye |  |  |  |  |  | -3.70 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 1 | 1
  Change From Baseline at Month 24: Study Eye |  |  |  |  | -6.28 (NA) — SD cannot be estimated for 1 participant. | -5.36 (NA) — SD cannot be estimated for 1 participant.
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 0 | 0 | 0 | 0 | 0 | 1
  Change From Baseline at Month 24: Non-Study Eye |  |  |  |  |  | -7.87 (NA) — SD cannot be estimated for 1 participant.

31. Secondary Outcome: Part 1: Change From Baseline in Contrast Sensitivity (CS) Score
Description: Change in CS was assessed by Pelli-Robson chart which uses a single large letter size (20/60 optotype), with contrast varying across groups of letters. Chart uses letters (6 per line), arranged in groups whose contrast varies from high to low. Participants read the letters, starting with the highest contrast, until they were unable to read two or three letters in a single group. Each group had three letters of the same contrast level, so there were three trials per contrast level. Participant is assigned a score based on the contrast of the last group in which two or three letters were correctly read. Score is a measure of the participant's log contrast sensitivity ranging from 0-2.25, with 0 being no letters read, and 2.25 being all letters read. Total CS score = [(total letters correct - 3) x 0.05].
Time Frame: Baseline, Months 3, 6, 12, and 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on scale
Units Other Than Participants: eyes
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Number analyzed (eyes) | 6 | 6 | 6 | 6 | 6 | 6
Score on scale
  Baseline: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Study Eye | 0.300 (0.1732) | 0.533 (0.2309) | 0.900 (0.1732) | 0.883 (0.3884) | 1.267 (0.0289) | 1.067 (0.6110)
  Baseline: Non-Study: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Baseline: Non-Study | 0.433 (0.2082) | 0.583 (0.2255) | 1.050 (0.2598) | 0.933 (0.4646) | 1.350 (0.1803) | 1.100 (0.3279)
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Study Eye | 0.167 (0.1528) | 0.183 (0.2566) | 0.150 (0.0866) | 0.133 (0.1155) | -0.033 (0.4163) | -0.167 (0.3014)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 3: Non-Study Eye | 0.000 (0.0000) | 0.017 (0.4010) | 0.050 (0.0500) | 0.050 (0.0500) | 0.100 (0.0000) | 0.000 (0.1000)
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Study Eye | 0.133 (0.2082) | 0.067 (0.2363) | 0.100 (0.1323) | 0.133 (0.0577) | -0.183 (0.4072) | 0.117 (0.2021)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 6: Non-Study Eye | 0.000 (0.1732) | 0.033 (0.2255) | 0.083 (0.0764) | 0.050 (0.1000) | -0.100 (0.0500) | 0.000 (0.0500)
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Study Eye | 0.100 (0.2828) | 0.133 (0.3512) | -0.017 (0.1041) | 0.183 (0.0577) | -0.167 (0.6788) | -0.017 (0.3329)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 12: Non-Study Eye | -0.100 (0.2828) | 0.067 (0.3512) | 0.000 (0.0000) | 0.000 (0.0500) | -0.100 (0.1323) | -0.050 (0.1323)
  Change From Baseline at Month 24: Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Study Eye | 0.000 (0.2291) | 0.017 (0.5965) | -0.100 (0.0000) | 0.217 (0.1893) | -0.217 (0.5346) | -0.117 (0.2466)
  Change From Baseline at Month 24: Non-Study Eye: number analyzed (eyes) | 3 | 3 | 3 | 3 | 3 | 3
  Change From Baseline at Month 24: Non-Study Eye | -0.183 (0.1258) | 0.117 (0.3884) | -0.100 (0.1732) | 0.017 (0.2021) | -0.050 (0.1323) | 0.050 (0.0500)

32. Secondary Outcome: Part 2: Percentage of Study Eyes With ≥7 dB Improvement From Baseline at ≥5 Points Out of the 16 Central Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dBs using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' is assigned a value of '-1' by MAIA in the calculation. Improvement in mean sensitivity in center grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points out of the 16 central points.
Time Frame: Months 1, 2, 3, 6, and 9
Population: ITT analysis set included all participants who were randomized, under the 3-arm randomization schedules. 'Number analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Number (80% Confidence Interval); unit: percentage of study eyes
Units Other Than Participants: study eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (study eyes) | 9 | 10 | 10
percentage of study eyes
  Month 1 | 22.2 [6.1 to 49.0] | 30.0 [11.6 to 55.2] | 40.0 [18.8 to 64.6]
  Month 2 | 22.2 [6.1 to 49.0] | 30.0 [11.6 to 55.2] | 50.0 [26.7 to 73.3]
  Month 3: number analyzed (Participants) | 8 | 10 | 10
  Month 3: number analyzed (study eyes) | 8 | 10 | 10
  Month 3 | 12.5 [1.3 to 40.6] | 30.0 [11.6 to 55.2] | 60.0 [35.4 to 81.2]
  Month 6: number analyzed (Participants) | 9 | 9 | 8
  Month 6: number analyzed (study eyes) | 9 | 9 | 8
  Month 6 | 22.2 [6.1 to 49.0] | 33.3 [12.9 to 59.9] | 62.5 [34.5 to 85.3]
  Month 9: number analyzed (Participants) | 9 | 7 | 7
  Month 9: number analyzed (study eyes) | 9 | 7 | 7
  Month 9 | 22.2 [6.1 to 49.0] | 28.6 [7.9 to 59.6] | 42.9 [17.0 to 72.1]

33. Secondary Outcome: Part 2: Percentage of Study Eyes With ≥7 dB Improvement From Baseline at ≥5 Points Out of the 68 Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dBs using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Improvement in mean sensitivity in whole grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points of the grid as a whole (68 points).
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 32
Measure: Number (80% Confidence Interval); unit: percentage of study eyes
Units Other Than Participants: study eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (study eyes) | 9 | 10 | 10
percentage of study eyes
  Month 1 | 33.3 [12.9 to 59.9] | 60.0 [35.4 to 81.2] | 40.0 [18.8 to 64.6]
  Month 2 | 22.2 [6.1 to 49.0] | 80.0 [55.0 to 94.5] | 80.0 [55.0 to 94.5]
  Month 3 | 25.0 [6.9 to 53.8] | 80.0 [55.0 to 94.5] | 70.0 [44.8 to 88.4]
  Month 6 | 33.3 [12.9 to 59.9] | 77.8 [51.0 to 93.9] | 100.0 [75.0 to 100.0]
  Month 9 | 33.3 [12.9 to 59.9] | 85.7 [54.7 to 98.5] | 71.4 [40.4 to 92.1]
  Month 12 | 33.3 [12.9 to 59.9] | 62.5 [34.5 to 85.3] | 62.5 [34.5 to 85.3]

34. Secondary Outcome: Part 2: Change From Baseline in Mean Sensitivity of the 16 Central Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Mean Sensitivity in center grid was defined as the mean in dB of the 16 points located in the center of the grid. Here negative values indicate a decline in retinal sensitivity.
Time Frame: Baseline, Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
dBs
  Baseline: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Study Eye | 6.78 (3.488) | 7.39 (5.207) | 7.38 (3.095)
  Baseline: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Non-Study Eye | 9.56 (3.321) | 9.09 (5.003) | 8.98 (3.583)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Study Eye | 1.53 (3.086) | 2.70 (3.731) | 0.10 (5.723)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Non-Study Eye | -0.26 (1.692) | -0.76 (1.793) | -0.08 (0.834)
  Change From Baseline at Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Study Eye | 1.62 (2.846) | 2.73 (4.360) | 1.55 (5.886)
  Change From Baseline at Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Non-Study Eye | -0.34 (2.027) | -0.44 (1.723) | 0.26 (1.118)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye | 1.17 (2.760) | 2.77 (4.598) | 1.00 (6.862)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | -1.24 (1.253) | 0.07 (1.393) | -0.24 (0.500)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye | 0.72 (3.208) | 3.38 (4.770) | 3.74 (3.931)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | -0.69 (2.199) | -0.35 (1.125) | -0.66 (0.702)
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 9 | 7 | 7
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 9 | 7 | 7
  Change From Baseline at Month 9: Study Eye | 0.65 (3.272) | 2.52 (4.619) | 2.54 (6.317)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye | -1.01 (1.943) | 0.30 (1.654) | -0.54 (0.636)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 9 | 8 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 9 | 8 | 8
  Change From Baseline at Month 12: Study Eye | -0.11 (4.446) | 2.79 (4.663) | 1.16 (5.660)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye | -2.23 (4.018) | -0.44 (1.078) | -1.04 (1.292)

35. Secondary Outcome: Part 2: Change From Baseline in Mean Sensitivity of the 68 Central Loci Points of the 10-2 Grid Assessed by MAIA Microperimetry
Description: MAIA microperimetry assessment was measured in dB using a 10-2 grid of 68 points. Each point was labelled as '< 0', '0' or a positive integer. The point labelled as '< 0' was assigned a value of '-1' by MAIA in the calculation. Improvement in mean ensitivity in whole grid was defined as an increase from baseline of 7 or more dBs in any 5 or more points of the grid as a whole (68 points). Here negative values indicate a decline in retinal sensitivity.
Time Frame: Baseline, Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
dBs
  Baseline: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Study Eye | 2.15 (2.182) | 2.46 (1.911) | 3.84 (2.138)
  Baseline: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Non-Study Eye | 3.32 (2.539) | 3.34 (2.092) | 4.47 (2.331)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Study Eye | 0.91 (1.389) | 1.60 (2.225) | -0.07 (3.898)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Non-Study Eye | 0.12 (1.214) | -0.46 (1.044) | -0.03 (0.850)
  Change From Baseline at Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Study Eye | 0.90 (0.972) | 2.34 (2.353) | 1.18 (3.367)
  Change From Baseline at Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Non-Study Eye | 0.30 (1.111) | -0.23 (0.859) | 0.13 (0.668)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye | 0.46 (1.064) | 2.64 (2.962) | 0.24 (3.962)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | -0.16 (0.743) | -0.03 (0.516) | -0.11 (0.619)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye | 0.32 (1.301) | 3.15 (3.283) | 2.05 (3.007)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | -0.13 (1.283) | -0.27 (0.527) | -0.50 (0.632)
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 9 | 7 | 7
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 9 | 7 | 7
  Change From Baseline at Month 9: Study Eye | 0.40 (1.456) | 2.80 (3.116) | 1.71 (3.605)
  Change From Baseline at Month 9: Non- Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Non- Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Non- Study Eye | -0.41 (1.150) | -0.05 (0.790) | 0.09 (0.544)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 9 | 8 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 9 | 8 | 8
  Change From Baseline at Month 12: Study Eye | 0.11 (1.592) | 2.79 (3.045) | 0.89 (3.132)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye | -0.84 (1.749) | -0.28 (0.476) | -0.35 (1.004)

36. Secondary Outcome: Part 2: Change From Baseline in BCVA Reported as Letters
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. BCVA was reported as number of letters read correctly by the participant, using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate a decline in BCVA.
Time Frame: Baseline, Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
letters
  Baseline: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Study Eye | 68.78 (5.954) | 65.90 (10.104) | 68.20 (8.991)
  Baseline: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Non-Study Eye | 72.89 (6.846) | 68.50 (9.675) | 68.80 (6.989)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Study Eye | 0.44 (2.833) | 1.60 (6.450) | 0.60 (7.545)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Non-Study Eye | -0.89 (2.028) | 0.00 (4.110) | 3.80 (3.360)
  Change From Baseline at Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Study Eye | 0.22 (2.108) | -1.00 (12.392) | 0.00 (8.957)
  Change From Baseline at Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 2: Non-Study Eye | -0.11 (1.269) | 0.60 (2.836) | 3.10 (2.644)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye | 1.38 (2.615) | 0.10 (6.540) | -0.30 (11.036)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | 0.13 (2.642) | 1.10 (2.470) | 3.20 (2.860)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye | 1.00 (2.000) | 2.44 (5.003) | -0.38 (5.630)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | -1.56 (2.833) | 0.67 (1.581) | 1.00 (4.629)
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Study Eye | 0.44 (1.944) | -2.50 (14.263) | -0.57 (1.397)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye | -1.78 (2.949) | 1.00 (2.000) | 1.71 (3.147)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 12: Study Eye | 0.22 (2.949) | -4.00 (17.436) | -0.75 (3.370)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 7
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 7
  Change From Baseline at Month 12: Non-Study Eye | -4.11 (3.983) | 0.89 (3.100) | 2.14 (3.976)

37. Secondary Outcome: Part 2: Change From Baseline in Mean LLVA Reported as Letters
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. LLVA was reported as number of letters read correctly by the participant, using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate a decline in LLVA.
Time Frame: Baseline, Months 1, 3, 6, 9, and 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
letters
  Baseline: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Study Eye | 50.22 (13.349) | 39.30 (22.246) | 47.90 (14.970)
  Baseline: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Baseline: Non-Study Eye | 54.78 (11.872) | 49.50 (19.127) | 51.60 (9.524)
  Change From Baseline at Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Study Eye | 0.56 (7.618) | 11.30 (16.918) | -1.30 (18.397)
  Change From Baseline at Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Change From Baseline at Month 1: Non-Study Eye | 0.22 (5.215) | -3.00 (9.165) | 3.50 (4.882)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Study Eye | 3.63 (7.230) | 8.10 (16.251) | -3.50 (22.609)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | -0.63 (8.158) | 0.50 (3.749) | 1.20 (3.553)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Study Eye | 1.22 (7.032) | 8.00 (18.581) | 3.25 (14.636)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | 0.11 (6.274) | -3.56 (8.472) | 2.13 (2.850)
  Change From Baseline at Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Study Eye | -1.78 (7.225) | 8.38 (16.088) | 6.00 (12.356)
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Change From Baseline at Month 9: Non-Study Eye | -3.11 (7.491) | -1.13 (6.749) | 4.00 (4.082)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 12: Study Eye | -2.22 (7.412) | 5.11 (14.426) | -0.63 (11.575)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Change From Baseline at Month 12: Non-Study Eye | -4.44 (7.002) | -3.56 (11.652) | -1.50 (4.309)

38. Secondary Outcome: Part 2: Percentage of Eyes With a ≥15 Letter Increase From Baseline for BCVA
Description: as for outcome 11
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: ITT analysis set included all participants that were randomized under the 3-arm randomization schedules. 'Number analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7]
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 25.0]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 28.0]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 28.0]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 7
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 7
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 28.0]

39. Secondary Outcome: Part 2: Percentage of Eyes With a ≥15 Letter Increase From Baseline for LLVA
Description: as for outcome 12
Time Frame: Months 1, 3, 6, 9, and 12
Population: ITT analysis set included all participants that were randomized under the 3-arm randomization schedules. "Number analyzed" signifies the number of participants with data available for analysis at specified timepoint.
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 40.0 [18.8 to 64.6] | 20.0 [5.5 to 45.0]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 22.6] | 40.0 [18.8 to 64.6] | 30.0 [11.6 to 55.2]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 33.3 [12.9 to 59.9] | 12.5 [1.3 to 40.6]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 25.0]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 25.0 [6.9 to 53.8] | 28.6 [7.9 to 59.6]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 28.0]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 33.3 [12.9 to 59.9] | 12.5 [1.3 to 40.6]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0]

40. Secondary Outcome: Part 2: Percentage of Eyes With a ≥10 Letter Increase From Baseline for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Percentage of eyes with a ≥10 letters increase from baseline for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 20.0 [5.5 to 45.0]
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 3: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 12.5 [1.3 to 40.6]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 28.0]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 28.0]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 25.0]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 7
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 7
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 28.0]

41. Secondary Outcome: Part 2: Percentage of Eyes With a ≥10 Letter Increase From Baseline for LLVA
Description: as for outcome 14
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 11.1 [1.2 to 36.8] | 40.0 [18.8 to 64.6] | 30.0 [11.6 to 55.2]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 25.0 [6.9 to 53.8] | 40.0 [18.8 to 64.6] | 30.0 [11.6 to 55.2]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 12.5 [1.3 to 40.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 11.1 [1.2 to 36.8] | 44.4 [21.0 to 69.9] | 14.7 [14.7 to 65.5]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 11.1 [1.2 to 36.8] | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 25.0]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 11.1 [1.2 to 36.8] | 37.5 [14.7 to 65.5] | 28.6 [7.9 to 59.6]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 11.1 [1.2 to 36.8] | 12.5 [1.3 to 40.6] | 14.3 [1.5 to 45.3]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 11.1 [1.2 to 36.8] | 33.3 [12.9 to 59.9] | 12.5 [1.3 to 40.6]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 25.0]

42. Secondary Outcome: Part 2: Percentage of Eyes With a ≥5 Letter Increase From Baseline for BCVA
Description: as for outcome 15
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 60.0 [35.4 to 81.2] | 20.0 [5.5 to 45.0]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 40.0 [18.8 to 64.6]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 60.0 [35.4 to 81.2] | 30.0 [11.6 to 55.2]
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 30.0 [11.6 to 55.2]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 12.5 [1.3 to 40.6] | 20.0 [5.5 to 45.0] | 30.0 [11.6 to 55.2]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 20.6] | 20.0 [5.5 to 45.0]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 11.1 [1.2 to 36.8] | 44.4 [21.0 to 69.9] | 12.5 [1.3 to 40.6]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 25.0 [6.9 to 53.8]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 37.5 [14.7 to 65.5] | 0.0 [0.0 to 28.0]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 25.0] | 42.9 [17.0 to 72.1]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 22.2 [6.1 to 49.0] | 0.0 [0.0 to 25.0]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 7
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 7
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 28.6 [7.9 to 59.6]

43. Secondary Outcome: Part 2: Percentage of Eyes With a ≥5 Letter Increase From Baseline for LLVA
Description: as for outcome 16
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 22.2 [6.1 to 49.0] | 60.0 [35.4 to 81.2] | 40.0 [18.8 to 64.6]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 22.2 [6.1 to 49.0] | 30.0 [11.6 to 55.2] | 30.0 [11.6 to 55.2]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 37.5 [14.7 to 65.5] | 50.0 [26.7 to 73.3] | 30.0 [11.6 to 55.2]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 25.0 [25.0 to 53.8] | 20.0 [5.5 to 45.0] | 10.0 [1.0 to 33.7]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 44.4 [21.0 to 69.9] | 66.7 [40.1 to 87.1] | 50.0 [24.0 to 76.0]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 22.2 [6.1 to 49.0] | 11.1 [1.2 to 36.8] | 25.0 [6.9 to 53.8]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 22.2 [6.1 to 49.0] | 62.5 [34.5 to 85.3] | 57.1 [27.9 to 83.0]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 11.1 [1.2 to 36.8] | 12.5 [1.3 to 40.6] | 42.9 [17.0 to 72.1]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 22.2 [6.1 to 49.0] | 44.4 [21.0 to 69.9] | 12.5 [1.3 to 40.6]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Non-Study Eye | 11.1 [1.2 to 36.8] | 22.2 [6.1 to 49.0] | 0.0 [0.0 to 25.0]

44. Secondary Outcome: Part 2: Percentage of Eyes With a ≥15 Letters Loss From Baseline for BCVA
Description: as for outcome 21
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Part 2: Untreated Group: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 1 (5 × 10^9 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
- Part 2: BIIB112 Low Dose: Followed by vitrectomy and retinal detachment in the study eye, participants received a single dose 2 (1 × 10^10 vg) of BIIB112 by sub-retinal injection on Day 0 (surgery day).
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 18.9] | 8.3 [0.9 to 28.7]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]
  Month 2: Non- Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non- Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 18.9] | 8.3 [0.9 to 28.7]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 11.1 [1.2 to 36.8]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 10 | 9
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 9
  Month 12: Non-Study Eye | 0.0 [0.0 to 222.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 22.6]

45. Secondary Outcome: Part 2: Percentage of Eyes With a ≥15 Letters Loss From Baseline for LLVA
Description: as for outcome 18
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 18.9] | 33.3 [15.4 to 55.9]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 18.2 [4.9 to 41.5] | 0.0 [0.0 to 17.5]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 9.1 [1.0 to 31.0] | 33.3 [15.4 to 55.9]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 20.0 [5.5 to 45.0]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 11.1 [1.2 to 36.8]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 20.0 [5.5 to 45.0]
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Non-Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]

46. Secondary Outcome: Part 2: Percentage of Eyes With a ≥10 Letters Loss From Baseline for BCVA
Description: as for outcome 19
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 0.0 [0.0 to 22.6] | 9.1 [1.0 to 31.0] | 8.3 [0.9 to 28.7]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 10.0 [1.0 to 33.7]
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 9.1 [1.0 to 31.0] | 8.3 [0.9 to 28.7]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 0.0 [0.0 to 22.6] | 11.1 [1.2 to 36.8] | 11.1 [1.2 to 36.8]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 10.0 [1.0 to 33.7]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 10 | 9
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 9
  Month 12: Non-Study Eye | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 22.6]

47. Secondary Outcome: Part 2: Percentage of Eyes With a ≥10 Letters Loss From Baseline for LLVA
Description: as for outcome 20
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 18.9] | 33.3 [15.4 to 55.9]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 0.0 [0.0 to 22.6] | 18.2 [4.9 to 41.5] | 0.0 [0.0 to 17.5]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 18.2 [4.9 to 41.5] | 33.3 [15.4 to 55.9]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 12.5 [1.3 to 40.6] | 0.0 [0.0 to 18.9] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 20.0 [5.5 to 45.0]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 0.0 [0.0 to 20.6]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 11.1 [1.2 to 22.6] | 11.1 [1.2 to 36.8] | 11.1 [1.2 to 36.8]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 11.1 [1.2 to 36.8] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 30.0 [11.6 to 55.2]
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Non-Study Eye | 33.3 [12.9 to 59.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]

48. Secondary Outcome: Part 2: Percentage of Eyes With a ≥5 Letters Loss From Baseline for BCVA
Description: as for outcome 21
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 11.1 [1.2 to 36.8] | 9.1 [1.0 to 31.0] | 33.3 [15.4 to 55.9]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 11.1 [1.2 to 36.8] | 9.1 [1.0 to 31.0] | 0.0 [0.0 to 17.5]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 0.0 [0.0 to 22.6] | 20.0 [5.5 to 45.0] | 40.0 [18.8 to 64.6]
  Month 2: Non-Study Eye: number analyzed (Participants) | 9 | 10 | 9
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 9
  Month 2: Non-Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 20.6]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 0.0 [0.0 to 25.0] | 18.2 [4.9 to 41.5] | 33.3 [15.4 to 55.9]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 0.0 [0.0 to 25.0] | 18.2 [4.9 to 41.5] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 0.0 [0.0 to 22.6] | 10.0 [1.0 to 33.7] | 30.0 [11.6 to 55.2]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 22.2 [6.1 to 49.0] | 0.0 [0.0 to 20.6] | 10.0 [1.0 to 33.7]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 22.2 [6.1 to 49.0] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 22.2 [6.1 to 49.0] | 0.0 [0.0 to 22.6] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 11.1 [1.2 to 36.8] | 20.0 [5.5 to 22.6] | 20.0 [5.5 to 45.0]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 10 | 9
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 9
  Month 12: Non-Study Eye | 33.3 [12.9 to 59.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 22.6]

49. Secondary Outcome: Part 2: Percentage of Eyes With a ≥5 Letters Loss From Baseline for LLVA
Description: as for outcome 22
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 33.3 [12.9 to 59.9] | 18.2 [4.9 to 41.5] | 41.7 [21.9 to 63.8]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 33.3 [12.9 to 59.9] | 36.4 [16.9 to 59.9] | 0.0 [0.0 to 17.5]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 12.5 [1.3 to 40.6] | 18.2 [4.9 to 41.5] | 41.7 [21.9 to 63.8]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 37.5 [14.7 to 65.5] | 9.1 [1.0 to 31.0] | 0.0 [0.0 to 17.5]
  Month 6: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Study Eye | 22.2 [6.1 to 49.0] | 20.0 [5.5 to 45.0] | 30.0 [11.6 to 55.2]
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 6: Non-Study Eye | 33.3 [12.9 to 59.9] | 50.0 [26.7 to 73.3] | 0.0 [0.0 to 20.6]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Study Eye | 33.3 [12.9 to 59.9] | 22.2 [6.1 to 49.0] | 33.3 [12.9 to 59.9]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 9
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 9
  Month 9: Non-Study Eye | 55.6 [30.1 to 79.0] | 33.3 [12.9 to 59.9] | 0.0 [0.0 to 22.6]
  Month 12: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Study Eye | 55.6 [30.1 to 79.0] | 30.0 [11.6 to 55.2] | 40.0 [18.8 to 64.6]
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 12: Non-Study Eye | 44.4 [21.0 to 69.9] | 40.0 [18.8 to 64.6] | 30.0 [11.6 to 55.2]

50. Secondary Outcome: Part 2: Percentage of Eyes With Change From Baseline >-5 Letters for BCVA
Description: BCVA was assessed for both eyes using the ETDRS VA chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a change from baseline of ≥ -5 letters for BCVA were reported for study and non-study eyes.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 88.9 [63.2 to 98.8] | 90.0 [66.3 to 99.0] | 70.0 [44.8 to 88.4]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 88.9 [63.2 to 98.8] | 90.0 [66.3 to 99.0] | 100.0 [79.4 to 100.0]
  Month 2: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Study Eye | 100.0 [77.4 to 100.0] | 80.0 [55.0 to 94.5] | 60.0 [35.4 to 81.2]
  Month 2: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 2: Non-Study Eye | 100.0 [77.4 to 100.0] | 90.0 [66.3 to 99.0] | 100.0 [79.4 to 100.0]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 100.0 [75.0 to 100.0] | 80.0 [55.0 to 94.5] | 70.0 [44.8 to 88.4]
  Month 3: Non-Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Non-Study Eye | 100.0 [75.0 to 100.0] | 90.0 [66.3 to 99.0] | 100.0 [79.4 to 100.0]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 100.0 [77.4 to 100.0] | 88.9 [63.2 to 98.8] | 75.0 [46.2 to 93.1]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 77.8 [51.0 to 93.9] | 100.0 [77.4 to 100.0] | 87.5 [59.4 to 98.7]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 100.0 [77.4 to 100.0] | 75.0 [46.2 to 93.1] | 100.0 [72.0 to 100.0]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 77.8 [51.0 to 93.9] | 100.0 [75.0 to 100.0] | 100.0 [72.0 to 100.0]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 88.9 [63.2 to 98.8] | 77.8 [51.0 to 93.9] | 87.5 [59.4 to 98.7]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 7
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 7
  Month 12: Non-Study Eye | 66.7 [40.1 to 87.1] | 88.9 [63.2 to 98.8] | 100.0 [72.0 to 100.0]

51. Secondary Outcome: Part 2: Percentage of Eyes With Change From Baseline >-5 Letters for LLVA
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters were read at a distance of 4 meters from the chart. If <20 letters were read at 4 meters, testing at 1 meter was performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of eyes with a change from baseline of ≥ -5 letters for LLVA were reported for study and non-study eyes.
Time Frame: Months 1, 3, 6, 9, and 12
Population: as for outcome 38
Measure: Number (80% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (eyes) | 18 | 20 | 20
percentage of eyes
  Month 1: Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Study Eye | 66.7 [40.1 to 87.1] | 80.0 [55.0 to 94.5] | 70.0 [44.8 to 88.4]
  Month 1: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 1: Non-Study Eye | 66.7 [40.1 to 87.1] | 60.0 [35.4 to 81.2] | 100.0 [79.4 to 100.0]
  Month 3: Study Eye: number analyzed (Participants) | 8 | 10 | 10
  Month 3: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Month 3: Study Eye | 87.5 [59.4 to 98.7] | 80.0 [55.0 to 94.5] | 60.0 [35.4 to 81.2]
  Month 3: Non-Study Eye: number analyzed (eyes) | 9 | 10 | 10
  Month 3: Non-Study Eye | 62.5 [34.5 to 85.3] | 100.0 [79.4 to 100.0] | 100.0 [79.4 to 100.0]
  Month 6: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Study Eye | 77.8 [51.0 to 93.9] | 77.8 [51.0 to 93.9] | 75.0 [46.2 to 93.1]
  Month 6: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 6: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 6: Non-Study Eye | 66.7 [40.1 to 87.1] | 44.4 [21.0 to 69.9] | 100.0 [75.0 to 100.0]
  Month 9: Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Study Eye | 66.7 [40.1 to 87.1] | 75.0 [46.2 to 93.1] | 71.4 [40.4 to 92.1]
  Month 9: Non-Study Eye: number analyzed (Participants) | 9 | 8 | 7
  Month 9: Non-Study Eye: number analyzed (eyes) | 9 | 8 | 7
  Month 9: Non-Study Eye | 44.4 [21.0 to 69.9] | 62.5 [34.5 to 85.3] | 100.0 [72.0 to 100.0]
  Month 12: Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Study Eye | 44.4 [21.0 to 69.9] | 66.7 [40.1 to 87.1] | 75.0 [46.2 to 93.1]
  Month 12: Non-Study Eye: number analyzed (Participants) | 9 | 9 | 8
  Month 12: Non-Study Eye: number analyzed (eyes) | 9 | 9 | 8
  Month 12: Non-Study Eye | 55.6 [30.1 to 79.0] | 55.6 [30.1 to 79.0] | 62.5 [34.5 to 85.3]

52. Secondary Outcome: Part 2: Change From Baseline in Volume of 30-Degree Hill of Vision Assessed by Octopus 900
Description: Visual field testing was performed to assess the volume of 30-degree hill vision, reported as dBs. RF=number of false positive responses + number of false negative responses/number of false positive presentations + number of false negative presentations*100. If there are 0 responses, then RF value=0. RFpositive=number of false positive responses/number of false positive presentations*100. If RF≤ 20% measurement is considered reliable. If 20% < RF ≤ 25% and RFpositive ≤ 10% measurement is also considered reliable. Otherwise if 20% < RF ≤ 25% and RFpositive > 10%, or RF > 25%, measurement is not reliable. Only reliable measurements were included for analysis of this outcome measure. Here negative values indicate decline in the volume of 30-degree hill vision.
Time Frame: Baseline, Months 3, 6, and 12
Population: ITT analysis set included all participants that were randomized under the 3-arm randomization schedules. 'Overall number of participants analyzed' signifies the number of participants with data available for analysis of outcome measure. 'Number analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 8 | 10 | 10
Number analyzed (eyes) | 16 | 20 | 20
dBs
  Baseline: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Baseline: Study Eye | 3.61 (3.436) | 3.58 (2.549) | 5.70 (3.161)
  Baseline: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Baseline: Non-Study Eye | 3.05 (3.223) | 3.71 (2.668) | 6.23 (2.956)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 7 | 10 | 8
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 7 | 10 | 8
  Change From Baseline at Month 3: Study Eye | 0.80 (1.236) | 0.63 (1.162) | -0.01 (5.288)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 7 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 7 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | 0.52 (1.315) | 0.45 (0.759) | -0.02 (1.110)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 8 | 8 | 7
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 8 | 8 | 7
  Change From Baseline at Month 6: Study Eye | 0.13 (0.499) | 0.57 (1.354) | -1.22 (1.566)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 7 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 7 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | 0.20 (0.516) | 0.30 (0.665) | 0.19 (0.576)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 7 | 8 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 7 | 8 | 8
  Change From Baseline at Month 12: Study Eye | -0.36 (0.615) | 0.26 (1.164) | -1.91 (1.498)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 7 | 8 | 8
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 7 | 8 | 8
  Change From Baseline at Month 12: Non-Study Eye | 0.29 (0.487) | -0.10 (0.781) | -0.56 (0.337)

53. Secondary Outcome: Part 2: Change From Baseline in Volume of Full Field Hill of Vision Assessed by Octopus 900
Description: Visual field testing was performed to assess the volume of full field of hill vision, reported as dBs. RF=number of false positive responses + number of false negative responses/number of false positive presentations + number of false negative presentations*100. If there are 0 responses, then RF value=0. RFpositive=number of false positive responses/number of false positive presentations*100. If RF≤ 20% measurement is considered reliable. If 20% < RF ≤ 25% and RFpositive ≤ 10% measurement is also considered reliable. Otherwise if 20% < RF ≤ 25% and RFpositive > 10%, or RF > 25%, measurement is not reliable. Only reliable measurements were included for analysis of this outcome measure. Here negative values indicate decline in volume of full field hill vision.
Time Frame: Baseline, Months 3, 6, and 12
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: dBs
Units Other Than Participants: eyes
Arm/Group | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
Number analyzed (Participants) | 8 | 10 | 10
Number analyzed (eyes) | 16 | 20 | 20
dBs
  Baseline: Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Baseline: Study Eye | 7.26 (8.624) | 17.51 (17.302) | 19.48 (16.248)
  Baseline: Non-Study Eye: number analyzed (eyes) | 8 | 10 | 10
  Baseline: Non-Study Eye | 7.05 (8.821) | 16.33 (16.803) | 21.08 (17.560)
  Change From Baseline at Month 3: Study Eye: number analyzed (Participants) | 7 | 10 | 8
  Change From Baseline at Month 3: Study Eye: number analyzed (eyes) | 7 | 10 | 8
  Change From Baseline at Month 3: Study Eye | 1.84 (3.168) | 1.26 (3.327) | -0.10 (4.059)
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (Participants) | 7 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye: number analyzed (eyes) | 7 | 10 | 10
  Change From Baseline at Month 3: Non-Study Eye | 1.36 (2.460) | 2.01 (2.832) | 0.55 (3.097)
  Change From Baseline at Month 6: Study Eye: number analyzed (Participants) | 8 | 8 | 7
  Change From Baseline at Month 6: Study Eye: number analyzed (eyes) | 8 | 8 | 7
  Change From Baseline at Month 6: Study Eye | -0.35 (1.461) | 0.98 (2.197) | 1.52 (3.897)
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (Participants) | 7 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye: number analyzed (eyes) | 7 | 9 | 8
  Change From Baseline at Month 6: Non-Study Eye | 0.46 (1.124) | 0.99 (2.324) | 1.38 (2.526)
  Change From Baseline at Month 12: Study Eye: number analyzed (Participants) | 7 | 8 | 8
  Change From Baseline at Month 12: Study Eye: number analyzed (eyes) | 7 | 8 | 8
  Change From Baseline at Month 12: Study Eye | -1.18 (1.302) | 0.81 (3.709) | -0.95 (3.992)
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (Participants) | 7 | 8 | 8
  Change From Baseline at Month 12: Non-Study Eye: number analyzed (eyes) | 7 | 8 | 8
  Change From Baseline at Month 12: Non-Study Eye | 0.66 (1.193) | 0.28 (2.736) | -0.91 (2.001)

ADVERSE EVENTS:
Time Frame: Day 0 (surgery) in Part 1 of the study up to last follow up visit in Part 2 of the study (approximately 36 months)
Description: Safety analysis set consists of all participants who received study treatment (vitrectomy/BIIB112).
Arm/Group | Part 1: BIIB112 Dose 1 | Part 1: BIIB112 Dose 2 | Part 1: BIIB112 Dose 3 | Part 1: BIIB112 Dose 4 | Part 1: BIIB112 Dose 5 | Part 1: BIIB112 Dose 6 | Part 2: Untreated Group | Part 2: BIIB112 Low Dose | Part 2: BIIB112 High Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/9 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 0/3 | 1/3 | 2/3 | 1/9 | 3/11 | 5/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 5/9 | 11/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: BIIB112 Dose 1 (N=3) | Part 1: BIIB112 Dose 2 (N=3) | Part 1: BIIB112 Dose 3 (N=3) | Part 1: BIIB112 Dose 4 (N=3) | Part 1: BIIB112 Dose 5 (N=3) | Part 1: BIIB112 Dose 6 (N=3) | Part 2: Untreated Group (N=9) | Part 2: BIIB112 Low Dose (N=11) | Part 2: BIIB112 High Dose (N=12)
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Noninfective retinitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: BIIB112 Dose 1 (N=3) | Part 1: BIIB112 Dose 2 (N=3) | Part 1: BIIB112 Dose 3 (N=3) | Part 1: BIIB112 Dose 4 (N=3) | Part 1: BIIB112 Dose 5 (N=3) | Part 1: BIIB112 Dose 6 (N=3) | Part 2: Untreated Group (N=9) | Part 2: BIIB112 Low Dose (N=11) | Part 2: BIIB112 High Dose (N=12)
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraocular pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 6 | 5
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Visual field tests abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin d decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphotopsia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tunnel vision (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anterior chamber inflammation (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blindness transient (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 3
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Choroidal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 9
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Conjunctival irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal deposits (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Delayed light adaptation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyschromatopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hypotony of eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lenticular pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Noninfective retinitis (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 3
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Ocular hypertension (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal cyst (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal deposits (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Retinal fovea disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Retinal infiltrates (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Retinal thickening (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinoschisis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Vitreal cells (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypopyon (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aniseikonia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anterior chamber cell (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 6
Anterior chamber flare (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally, the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor's Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of the Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03116113/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03116113/SAP_001.pdf